CLINICAL TRIAL: NCT01661452
Title: Development of Post Traumatic Stress Disorder After Natural Disaster
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: F110510007
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Development of PTSD After Natural Disaster

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- patients in UAB ER,
  Interventions: Other: Referral to counseling services if desired

INTERVENTIONS:
Other: Referral to counseling services if desired

SUMMARY:
A survey (patient self-report) of patients presenting to UAB emergency room, outpatient trauma clinics and substance abuse center for symptoms of post-traumatic stress disorder and maladaptive coping responses after the widespread tornado disaster that occurred in Alabama in April 2011.

ELIGIBILITY:
Inclusion Criteria:

* 19 and older Able and willing to complete a questionnaire

Exclusion Criteria:

* Younger than 19 Unwilling or unable to complete a questionnaire

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to UAB emergency room, outpatient trauma clinics and substance abuse center.
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Development of PTSD | June 2011-December 2012

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States